CLINICAL TRIAL: NCT05288166
Title: CYCLONE 3: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Abemaciclib in Combination With Abiraterone Plus Prednisone in Men With High-Risk Metastatic Hormone-Sensitive Prostate Cancer
Brief Title: A Study of Abemaciclib (LY2835219) With Abiraterone in Men With Prostate Cancer That Has Spread to Other Parts of the Body and is Expected to Respond to Hormonal Treatment (Metastatic Hormone-Sensitive Prostate Cancer)
Acronym: CYCLONE 3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18448; I3Y-MC-JPEG (Other: Eli Lilly and Company); 2022-500461-28-06 (Other: EU Trial Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Prostatic Neoplasms; Neoplasm Metastasis; Urogenital Neoplasms; Physiological Effects of Drugs; Antineoplastic Agents; Antineoplastic Agents, Hormonal; Androgens; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Abiraterone Acetate; Steroid Synthesis Inhibitors; Cytochrome P-450; Enzyme Inhibitors; Prednisone; Prednisolone; Cyclin-Dependent Kinase 4; Cyclin-Dependent Kinase 6
Keywords: Metastatic Hormone Sensitive Prostate Cancer; mHSPC; Stage IV Prostate Cancer; Recurrent Prostate Cancer; De Novo Metastatic Prostate Cancer; High-Risk; Visceral metastasis; Cyclin-Dependent Kinase 4 (CDK4); Cyclin-Dependent Kinase 6 (CDK6); CDK4; CDK6; CDK4/6
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Urogenital Neoplasms | interventions — abemaciclib; abiraterone; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abemaciclib (Experimental): Participants received 200 milligram (mg) abemaciclib twice daily (BID) in combination with standard doses of 1000 mg abiraterone acetate once daily and 5mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
  Interventions: Drug: Abemaciclib; Drug: Abiraterone; Drug: Prednisone or Prednisolone
- Placebo (Active Comparator): Participants received placebo BID in combination with standard doses of 1000 mg abiraterone acetate once daily and 5mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
  Interventions: Drug: Abiraterone; Drug: Prednisone or Prednisolone; Drug: Placebo for Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Administered orally.
  Other Names: LY2835219
  Arms: Abemaciclib
Drug: Abiraterone — Administered orally.
Drug: Prednisone or Prednisolone — Administered orally.
Drug: Placebo for Abemaciclib — Administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn whether adding abemaciclib to abiraterone plus prednisone prolongs the time before prostate cancer gets worse. Participation may last approximately 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate (as the predominant histology)
* High-risk metastatic hormone-sensitive prostate cancer. High risk is defined as:

  * Greater than or equal to (≥)4 bone metastases by bone scan and/or
  * ≥1 visceral metastases by computed tomography or magnetic resonance imaging
* Must have initiated androgen deprivation therapy (ADT) with luteinizing hormone-releasing hormone (LHRH) agonist/antagonist or bilateral orchiectomy prior to randomization. Up to 3 months of ADT prior to randomization is permitted with or without first-generation anti-androgen.
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Prior treatment with abemaciclib or any other cyclin dependent kinase 4 and 6 (CDK4 & 6) inhibitor
* Development of metastatic prostate cancer in the context of castrate levels of testosterone
* Received any prior systemic therapy for metastatic prostate cancer (including investigational agents), except for ADT and first-generation anti-androgen
* Clinically significant cardiovascular disease as evidenced by myocardial infarction, arterial thrombotic events, or severe/unstable angina in the past 6 months, or New York Heart Association Class II to IV heart failure
* History of syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin, or sudden cardiac arrest. Chronic and hemodynamically stable atrial arrhythmia well-controlled on medical therapy is permitted
* Uncontrolled hypertension
* Clinically active or chronic liver disease, moderate/severe hepatic impairment
* Known untreated central nervous system (CNS) metastasis. Participants with a history of treated brain metastases are eligible if stable for at least 8 weeks prior to randomization and off corticosteroid for at least 2 weeks prior to randomization

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 925 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2027-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (266):
- United States (63):
  - Arizona Oncology Associates, P.C. - HOPE, Prescott, Arizona
  - Arizona Oncology Associates, P.C. - HOPE, Prescott Valley, Arizona
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Genesis Cancer and Blood Institute, Hot Springs, Arkansas
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - Providence Medical Foundation, Fullerton, California
  - Moores Cancer Center, La Jolla, California
  - MemorialCare Health System - Long Beach Medical Center, Long Beach, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - UCLA Hematology/Oncology - Santa Monica, Los Angeles, California
  - Torrance Memorial Physician Network / Cancer Care, Torrance, California
  - PIH Health Hematology Medical Oncology, Whittier, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - UCHealth Memorial Hospital, Colorado Springs, Colorado
  - UCHealth Harmony, Fort Collins, Colorado
  - Colorado West Healthcare System - Grand Valley Oncology, Grand Junction, Colorado
  - USO-Rocky Mountain Cancer Center, Littleton, Colorado
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Millennium Oncology Research Clinic, Hollywood, Florida
  - University of Miami Hospital and Clinics, Sylvester Cancer Center, Miami, Florida
  - Florida Cancer Specialist- East, West Palm Beach, Florida
  - Dwight D Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Summit Cancer Care DBA Candler Medical Oncology Practice, Savannah, Georgia
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - The University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky
  - Sarah Cannon Research Institute, Baton Rouge, Louisiana
  - Chesapeake Urology, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Reliant Medical Group, Worcester, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Minnesota Oncology/Hematology PA, Minneapolis, Minnesota
  - Care Access - Clifton, Clifton, New Jersey
  - Maimonides Cancer Center, Brooklyn, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Associated Medical Professionals - Urology, Syracuse, New York
  - Clinical Research Alliance, Westbury, New York
  - TriState Urologic Services PSC Inc., Cincinnati, Ohio
  - Northwest Cancer Specialist, Tigard, Oregon
  - MidLantic urology, Bala-Cynwyd, Pennsylvania
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Tennessee Oncology Chattanooga-SCRI, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Balcones, Austin, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Oncology - Carrollton, Flower Mound, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - USO - Texas Oncology Gulf Coast, Sugar Land, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - US Oncology Research Network, The Woodlands, Texas
  - Texas Oncology - Longview Cancer Center, Tyler, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - The University of Vermont Medical Center Inc., Burlington, Vermont
  - Oncology and Hematology Associates of Southwest Virginia Inc, Roanoke, Virginia
- Argentina (13):
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - Investigaciones Clinicas Moleculares (ICM), Buenos Aires, Buenos Aires F.D.
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires, Buenos Air
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Air
  - Fundación Cenit Para La Investigación En Neurociencias, CABA, Ciudad Autónoma de Buenos Aire
  - Centro Medico Privado CEMAIC, Capital, Córdoba Province
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Clinica Viedma, Viedma, Río Negro Province
  - Centro Medico San Roque, San Miguel de Tucumán, Tucumán Province
  - Centro Oncologico Korben, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Centro Urológico Profesor Bengió, Córdoba
  - Centro Polivalente de Asistencia e Investigacion Clinica - CER San Juan, San Juan
- Australia (18):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Macquarie University, Macquarie University, New South Wales
  - Icon Cancer Centre South Brisbane, South Brisbane, Queensland
  - Tasman Oncology Research, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Barwon Health, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
  - Epworth Freemasons, Richmond, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (4):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst, Oost-Vlaanderen
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Groeninge Campus Kennedylaan, Kortrijk, West-Vlaanderen
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
- Brazil (13):
  - Centro de Pesquisa Clínica do Instituto do Câncer do Ceará, Fortaleza, Ceará
  - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Centro Avançado de Tratamento Oncológico- CENANTRON, Belo Horizonte, Minas Gerais
  - Centro Integrado de Oncologia de Curitiba, Curitiba, Paraná
  - Hospital de Cancer de Londrina, Londrina, Paraná
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen, Santa Cruz do Sul, Rio Grande do Sul
  - Clínica de Oncologia Reichow, Blumenau, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Instituto de de Educação, pesquisa e Gestão em Saúde, Rio de Janeiro
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo, São Paulo
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- China (31):
  - Afflilated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Second Affiliated hospital of Anhui Medical University, Hefei, Anhui
  - Wannan Medical College Yijishan Hospital, Wuhu, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Centre, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Wuhan Union Hospital, Wuhan, Hubei
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Nanchong Central Hospital, Nanchong, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
- Czechia (8):
  - Nemocnice Horovice, Hořovice, Beroun
  - Masarykuv onkologicky ustav, Brno, Brno-město
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha 10
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Oblastni nemocnice Pribram, Příbram, Příbram
  - Fakultni Nemocnice u sv. Anny v Brne, Brno, South Moravian
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Urocentrum Praha, Prague
- France (11):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital Morvan, Brest, Brittany Region
  - Polyclinique De Blois, La Chaussée-Saint-Victor, Centre-Val de Loire
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - CHU Besançon, Besançon, Doubs
  - Centre de Cancérologie du Grand Montpellier, Montpellier, Languedoc-Roussillon
  - Hôpital privé du Confluent SAS, Nantes, Loire-Atlantique
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire-Atlantique
  - Institut Paoli-Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
  - Clinique Victor Hugo Le Mans, Le Mans, Sarthe
  - Hôpital Européen Georges Pompidou, Paris
- Germany (16):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - NCT, Heidelberg, Baden-Wurttemberg
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Würt
  - Klinikum Rechts Der Isar Der Technischen Universität München, Munich, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Urologicum Duisburg Fachärztesozietät - Walsum, Duisburg, North Rhine-Westphalia
  - Urologische Gemeinschaftspraxis Heinsberg, Heinsberg, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - Urologische Gemeinschaftspraxis Wesel, Wesel, North Rhine-Westphalia
  - InVO Institut für Versorgungsforschung in der Onkologie, Koblenz, Rhineland-Palatinate
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Urologie Neandertal - Praxis Mettmann, Mettmann
  - Klinikum Nürnberg Nord, Nuremberg
- Greece (5):
  - University Hospital of Patras, Pátrai, Achaḯa
  - Agios Savvas Regional Cancer Hospital, Athens, Attikí
  - Alexandra Hospital, Athens, Attikí
  - Attikon General University Hospital, Chaïdári, Attikí
  - University General Hospital of Heraklion, Heraklion, Irakleío
- Hungary (4):
  - Bacs-Kiskun Megyei Korhaz, Kecskemét, Bács-Kiskun county
  - Petz Aladar Egyetemi Oktato Korhaz, Győr, Győr-Moson-Sopron
  - Országos Onkológiai Intézet, Budapest, Pest County
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
- Israel (7):
  - Meir Medical Center, Kfar Saba, Central District
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Yitzhak Shamir Medical Center, Ẕerifin, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Sourasky Medical Center, Tel Aviv, Tell Abīb
- Italy (7):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Istituto Oncologico Veneto IRCCS, Castelfranco Veneto, Veneto
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Azienda Ospedaliera Santa Maria Terni, Terni
  - APSS- Presidio Ospedaliero S. Chiara, Trento
- Japan (15):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kimitsu Chuo Hospital, Kisarazu, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kita, Kagawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Nagano Municipal Hospital, Tomitake, Nagano
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Showa University Hospital, Shinagawa, Tokyo
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Osaka International Cancer Institute, Osaka
  - Osaka Metropolitan University Hospital, Osaka
- Mexico (6):
  - Actualidad Basada en la Investigación del Cáncer, Guadalajara, Jalisco
  - Health Pharma Professional Research S.A. de C.V:, Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán, Sinaloa
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
- Netherlands (2):
  - ETZ Elisabeth, Tilburg, North Brabant
  - University Medical Center Groningen, Groningen
- Poland (5):
  - Clinical Best Solutions, Lublin, Lublin Voivodeship
  - Opolskie Centrum Onkologii w Opolu im. prof. Tadeusza Koszarowskiego, Opole, Opole Voivodeship
  - Szpitale Pomorskie Sp. z o. o., Gdynia, Pomeranian Voivodeship
  - Salve Medica, Lodz, Łódź Voivodeship
  - Provita Profamilia, Piotrkow Trybunalski, Łódź Voivodeship
- Romania (8):
  - C.M.D.T.A. Neomed, Brasov, Brașov County
  - Amethyst Radiotherapy Center, Florești, Cluj
  - Ovidius Clinical Hospital OCH, Ovidiu, Constanța County
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Radiology Therapeutic Center, Otopeni, Ilfov
  - Oncopremium Team, Baia Mare, Maramureş
  - SC Memorial Healthcare International SRL, Bucharest
  - Gral Medical Diagnostic Center, Bucharest
- South Korea (4):
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (7):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, Hospitalet, Barcelona [Barcelona]
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Fundación Instituto Valenciano de Oncología, Valencia, Valenciana, Comunitat
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario Virgen Del Rocio, Seville
- Taiwan (6):
  - National Taiwan University Hospital, Taipei City, Taipei
  - Taipei Veterans General Hospital, Taipei City, Taipei
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (9):
  - Medipol Mega Universite Hastanesi, Stanbul, Istanbul
  - Izmir Medical Park Hospital, Izmir, Karsiyaka, İzmir
  - Baskent University Dr. Turgut Noyan Research and Training Center, Adana
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Dicle Üniversitesi, Diyarbakır
  - Trakya University, Edirne
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi, Malatya
- United Kingdom (3):
  - Royal Blackburn Hospital, Blackburn, Blackburn With Darwen
  - Colchester General Hospital, Colchester, Essex
  - University College London Hospital, London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Abemaciclib (LY2835219) With Abiraterone in Men With Prostate Cancer That Has Spread to Other Parts of the Body and is Expected to Respond to Hormonal Treatment (Metastatic Hormone-Sensitive Prostate Cancer) (CYCLONE 3) — https://trials.lillytrialguide.com/en-US/trial/23jmzMPWglYwUwUN2GWvdM

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who had an event (radiographic progression or death) and participants who were off the treatment and were alive at study conclusion.
Groups:
- Abemaciclib: Participants received 200 milligram (mg) abemaciclib twice daily (BID) in combination with standard doses of 1000 mg abiraterone acetate once daily and 5 mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
- Placebo: Participants received placebo BID in combination with standard doses of 1000 mg abiraterone once daily and 5 mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
Period: Overall Study
Arm/Group | Abemaciclib | Placebo
Started | 463 | 462
Received at Least One Dose of Study Drug | 460 | 460
Completed | 47 | 39
Not Completed | 416 | 423
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Screen Failure | 1 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — On Study Treatment | 408 | 418

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Abemaciclib: Participants received 200 mg abemaciclib BID in combination with standard doses of 1000 mg abiraterone acetate once daily and 5mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
- Total: Total of all reporting groups
Arm/Group | Abemaciclib | Placebo | Total
Number analyzed (Participants) | 463 | 462 | 925
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.80 (8.16) | 69.30 (8.07) | 69.00 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 463 | 462 | 925
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 115 | 126 | 241
  Not Hispanic or Latino | 276 | 271 | 547
  Unknown or Not Reported | 72 | 65 | 137
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 27 | 27 | 54
  Asian | 122 | 120 | 242
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 17 | 15 | 32
  White | 278 | 286 | 564
  More than one race | 9 | 5 | 14
  Unknown or Not Reported | 9 | 9 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 40 | 39 | 79
  Australia | 28 | 29 | 57
  Belgium | 3 | 0 | 3
  Brazil | 46 | 53 | 99
  Canada | 1 | 1 | 2
  China | 65 | 70 | 135
  Czechia | 15 | 11 | 26
  France | 14 | 9 | 23
  Germany | 24 | 22 | 46
  Greece | 2 | 4 | 6
  Hungary | 5 | 5 | 10
  Israel | 7 | 9 | 16
  Italy | 12 | 12 | 24
  Japan | 39 | 30 | 69
  Mexico | 34 | 34 | 68
  Netherlands | 2 | 5 | 7
  Poland | 12 | 14 | 26
  Romania | 3 | 2 | 5
  South Korea | 7 | 4 | 11
  Spain | 16 | 14 | 30
  Taiwan | 8 | 7 | 15
  Turkey | 21 | 20 | 41
  United Kingdom | 7 | 1 | 8
  United States | 52 | 67 | 119

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-Free Survival (rPFS) Assessed by Investigator
Description: The rPFS time is measured from the date of randomization to the earliest date of investigator determined radiographic disease progression (by objective radiographic disease assessment per response evaluation criteria in solid tumors (RECIST) version 1.1 for soft tissue AND/OR radionuclide bone scan using prostate cancer working group 3 -PCWG3 criteria for bone) or death from any cause, whichever occurs first.
Time Frame: From Date of Randomization to Radiographic Disease Progression or Death from Any Cause (up to 22 months)
Population: All randomized participants (including the censored participants). Number of participants censored in "Abemaciclib = 385," "Placebo = 389."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 463 | 462
Months | NA [NA to NA] — Due to high number of censored participants, the median, upper and lower limit 95% confidence interval were not estimable. | NA [NA to NA] — Due to high number of censored participants, the median, upper and lower limit 95% confidence interval were not estimable.

2. Secondary Outcome: Radiographic Progression-Free Survival (rPFS) Assessed by Blinded Independent Central Review (BICR)
Description: as for outcome 1
Time Frame: From Date of Randomization to Radiographic Disease Progression or Death from Any Cause (up to 22 months)
Population: All randomized participants (including the censored participants). Number of participants censored in "Abemaciclib = 435," "Placebo = 440"
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 463 | 462
Months | NA [11.11 to NA] — Due to high number of censored participants, the median, and upper limit of 95% confidence interval were not estimable. | NA [13.02 to NA] — Due to high number of censored participants, the median, and upper limit of 95% confidence interval were not estimable.

3. Secondary Outcome: Castration-resistant Prostate Cancer (CRPC)-Free Survival
Description: CRPC-free survival is defined as the time from the date of randomization to the earliest date of castration resistance, as demonstrated by any of the following (whichever occurs earliest):
  Confirmed prostate-specific antigen (PSA) progression with serum testosterone ≤50 nanogram/deciliter (ng/dL) (≤1.73 nanomoles per liter(nmol/L)).
  Investigator-assessed radiographic progression with serum testosterone ≤50 ng/dL (≤1.73 nmol/L).
  Death from any cause.
Time Frame: Randomization to the earliest date of PSA or radiographic progression with a testosterone level of ≤50 ng/dL; or death from any cause (up to 22 months)
Population: All randomized participants (including the censored participants). Number of participants censored in "Abemaciclib = 363," "Placebo = 360."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 463 | 462
Months | NA [14.86 to NA] — Due to high number of censored participants, the median, upper limit of 95% confidence interval was not estimable. | NA [NA to NA] — Due to high number of censored participants, the median, upper and lower limit 95% confidence interval were not estimable.

4. Secondary Outcome: Overall Survival (OS)
Description: The OS time is measured from the date of randomization to the date of death from any cause. If the participant was alive or lost to follow-up at the time of data analysis, OS data were censored on the last date the participant was known to be alive.
Time Frame: From Date of Randomization to Date of Death Due to Any Cause (Up to 22 Months)
Population: All randomized participants (including the censored participants). Number of participants censored in "Abemaciclib = 416," "Placebo = 430."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 463 | 462
Months | NA [NA to NA] — Due to high number of censored participants, the median, upper and lower limit 95% confidence interval were not estimable. | NA [NA to NA] — Due to high number of censored participants, the median, upper and lower limit 95% confidence interval were not estimable.

5. Secondary Outcome: Time to Pain Progression
Time Frame: Randomization to pain progression (up to 22 months)
Population: All randomized participants (including the censored participants). Number of participants censored in "Abemaciclib = 368," "Placebo = 343"
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 463 | 462
Months | NA [NA to NA] — Due to high number of censored participants, the median, upper and lower limit of 95% confidence interval were not estimable. | 19.13 [15.35 to NA] — Due to high number of censored participants, the upper limit of 95% confidence interval was not estimable.

6. Secondary Outcome: Time to Deterioration in Health-Related Quality of Life (HRQoL) Measured by Functional Assessment of Cancer Therapy-Prostate (FACT-P) - Physical Well-Being Subscale
Description: Time to deterioration in health-related quality of life (HRQoL) was defined as the time from randomization to the date of the first clinically meaningful HRQoL deterioration on 2 consecutive measurements. HRQoL evaluation was performed using the FACT-P questionnaire. Physical Well-Being subscale is a subsection of FACT-P questionnaire. FACT-P consists of 39 core items to assess health related quality of life in participants with prostate cancer. It consisted of 5 sub-scales assessing physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and prostate cancer subscale (12 items). Each item is rated from 0 (Not at all) to 4 (Very much) and combined to produce subscale scores. FACT-P total score was the sum of all 5 subscale scores. It ranged from 0 to 156 with higher score indicating better quality of life. Physical well-being subscale score ranges from 0 to 28 with high score indicating better quality of life.
Time Frame: Randomization to the date of the first clinically meaningful HRQoL deterioration (up to 22 months)
Population: All randomized participants (including the censored participants). Number of participants censored in "Abemaciclib = 328," "Placebo = 394"
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 463 | 462
Months | NA [NA to NA] — Due to high number of censored participants, the median, upper and lower limit of 95% confidence interval were not estimable. | NA [NA to NA] — Due to high number of censored participants, the median, upper and lower limit of 95% confidence interval were not estimable.

7. Secondary Outcome: Time to Deterioration in Health-Related Quality of Life (HRQoL) Measured by Functional Assessment of Cancer Therapy-Prostate (FACT-P) - Prostate Cancer Subscale
Description: Time to deterioration in health-related quality of life (HRQoL) was defined as the time from randomization to the date of the first clinically meaningful HRQoL deterioration on 2 consecutive measurements. HRQoL evaluation was performed using the FACT-P questionnaire. Prostate Cancer Subscale is a subsection of FACT-P questionnaire. FACT-P consists of 39 core items to assess health related quality of life in participants with prostate cancer. It consisted of 5 sub-scales assessing physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and prostate cancer subscale (12 items). Each item is rated from 0 (Not at all) to 4 (Very much) and combined to produce subscale scores. FACT-P total score was the sum of all 5 subscale scores. It ranged from 0 to 156 with higher score indicating better quality of life. Prostate cancer subscale score ranges from 0 to 48 with high score indicating better quality of life.
Time Frame: Randomization to the date of the first clinically meaningful HRQoL deterioration (up to 22 months)
Population: All randomized participants (including the censored participants). Number of participants censored in "Abemaciclib = 329," "Placebo = 365."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 463 | 462
Months | NA [NA to NA] — Due to high number of censored participants, the median, upper and lower limit of 95% confidence interval were not estimable. | NA [NA to NA] — Due to high number of censored participants, the median, upper and lower limit of 95% confidence interval were not estimable.

8. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration at Steady State (Cmax,ss) of Abemaciclib
Description: Maximum plasma concentration at steady state (Cmax,ss) of abemaciclib was evaluated.
Time Frame: Predose on Cycle 1 Day 1, Predose and Predose on Cycle 2 Day 1 and Predose on Cycle 3 Day 1 (28 Day Cycles)
Population: All randomized participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Abemaciclib
Number analyzed (Participants) | 454
nanogram per milliliter (ng/mL) | 308.3 (50)

ADVERSE EVENTS:
Time Frame: Baseline up to 22 months
Description: All participants who received at least one dose of the study drug, regardless of their eligibility for the study.
Arm/Group | Abemaciclib | Placebo
All-Cause Mortality (participants affected / at risk) | 47/460 | 32/460
Serious Adverse Events (participants affected / at risk) | 145/460 | 68/460
Other Adverse Events (participants affected / at risk) | 445/460 | 380/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=460) | Placebo (N=460)
Anaemia (Blood and lymphatic system disorders) | 9 (10) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 5 (5) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 4 (4)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 3 (3)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Splenic artery aneurysm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 7 (7) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Stenosis (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 5 (5) | 3 (4)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 19 (20) | 4 (4)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (4) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 11 (13) | 3 (3)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Troponin t increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (9) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Perivascular epithelioid cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 8 (8) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (5) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Extrinsic iliac vein compression (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=460) | Placebo (N=460)
Anaemia (Blood and lymphatic system disorders) | 252 (317) | 58 (72)
Leukopenia (Blood and lymphatic system disorders) | 126 (259) | 10 (15)
Lymphopenia (Blood and lymphatic system disorders) | 45 (84) | 20 (29)
Neutropenia (Blood and lymphatic system disorders) | 217 (395) | 13 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 125 (198) | 14 (20)
Abdominal pain (Gastrointestinal disorders) | 73 (84) | 34 (40)
Constipation (Gastrointestinal disorders) | 45 (53) | 43 (51)
Diarrhoea (Gastrointestinal disorders) | 301 (636) | 62 (76)
Nausea (Gastrointestinal disorders) | 116 (150) | 41 (48)
Vomiting (Gastrointestinal disorders) | 65 (92) | 22 (25)
Fatigue (General disorders) | 178 (223) | 91 (102)
Malaise (General disorders) | 24 (29) | 8 (10)
Oedema peripheral (General disorders) | 66 (82) | 31 (40)
Pyrexia (General disorders) | 38 (45) | 14 (16)
Covid-19 (Infections and infestations) | 28 (29) | 21 (21)
Urinary tract infection (Infections and infestations) | 45 (56) | 22 (27)
Alanine aminotransferase increased (Investigations) | 63 (82) | 77 (93)
Aspartate aminotransferase increased (Investigations) | 53 (68) | 70 (87)
Blood alkaline phosphatase increased (Investigations) | 26 (30) | 15 (15)
Blood bilirubin increased (Investigations) | 25 (35) | 28 (53)
Blood creatinine increased (Investigations) | 130 (193) | 17 (22)
Weight decreased (Investigations) | 32 (37) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 87 (99) | 9 (10)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 25 (37) | 20 (25)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (19) | 31 (35)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 50 (62) | 47 (66)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25 (43) | 14 (23)
Hypokalaemia (Metabolism and nutrition disorders) | 133 (240) | 63 (106)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (36) | 39 (47)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (27) | 34 (43)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (21) | 25 (31)
Dizziness (Nervous system disorders) | 35 (43) | 24 (26)
Dysgeusia (Nervous system disorders) | 37 (41) | 4 (4)
Headache (Nervous system disorders) | 36 (40) | 34 (41)
Pollakiuria (Renal and urinary disorders) | 24 (26) | 19 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (47) | 35 (43)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 15 (17)
Rash (Skin and subcutaneous tissue disorders) | 42 (46) | 18 (19)
Hot flush (Vascular disorders) | 69 (74) | 98 (106)
Hypertension (Vascular disorders) | 52 (66) | 69 (76)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT05288166/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT05288166/SAP_001.pdf